CLINICAL TRIAL: NCT02181244
Title: Egg Effects on Atherogenic Dyslipidemia, Glucose Metabolism and Inflammation in Diabetic Subjects
Brief Title: Egg Effects on Atherogenic Dyslipidemias, Glucose Metabolism and Inflammation in Diabetic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H12-059
Record Dates: First submitted 2014-06-20; First posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus; Inflammation
Keywords: egg; oatmeal; atherogenic dyslipidemia; glycosylated hemoglobin; inflammatory markers
MeSH Terms: conditions — Diabetes Mellitus; Inflammation | interventions — Eggs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Egg, one a day, for breakfast (Experimental): The intervention consists in feeding the subjects egg, one a day for breakfast during 5 weeks. At the end of the intervention, blood will be obtained to measure plasma lipids, glucose, insulin and inflammatory markers. All measurements will be finished 24 weeks after the intervention is finished. All data will be reported 1 year after completion of the study.
  Interventions: Other: Egg, one a day, for breakfast; Other: Oatmeal, one cup a day
- Oatmeal, one cup a day (Experimental): In this arm, subjects will consume oatmeal for a period of 5 weeks. Blood samples will be taken and different parameters will be measured including plasma lipids, glucose, insulin and inflammatory markers. All these measurements will be finished 24 weeks after completion of the study. All data will be reported 1 year after completion of the study.
  Interventions: Other: Egg, one a day, for breakfast; Other: Oatmeal, one cup a day

INTERVENTIONS:
Other: Egg, one a day, for breakfast — One egg per day as breakfast for 5 weeks followed by a 3 week washout period and 5 additional weeks on oatmeal. This is a randomized crossover design. Half of subjects started with the eggs and the other half with oatmeal. Blood lipids, glucose and inflammatory measurements will be finished 24. weeks after completion of the study. Data will be reported 1 year after the completion of the study.
Other: Oatmeal, one cup a day — Subjects will be fed oatmeal for a period of 5 weeks. After 3 weeks they will be switched to the alternate diet. This is a randomized control trail in which plasma glucose, plasma lipids and inflammatory markers will be measured. All these measurements will be finished 24 weeks after completion of the study. Data will be reported after 1 year of the completion of the study.

SUMMARY:
There is concern in the literature regarding egg consumption in diabetic people. The investigators hypothesis is that compared to an oatmeal-based breakfast, an egg-based breakfast will not increase the risk for heart disease in diabetic people but it may reduce inflammation, in this population characterized by chronic low grade inflammation.

This is a cross-over study in which subjects will be randomly allocated to consume 1 egg per day for breakfast or a bowl of oatmeal with lactose-free milk for 5 weeks. After a 3 wk washout period, subjects will be allocated to the alternate treatment for additional 5 weeks.

Blood will be collected at baseline and at the end of each dietary period to measure plasma lipids, glucose, insulin, glycosylated hemoglobin and inflammatory markers.

DETAILED DESCRIPTION:
This study is conducted in diabetic patients who are given two distinct breakfasts: eggs and oatmeal in a crossover design. The investigators hypothesis is that eggs will not increase the risk for heart disease in this population when compared to oatmeal but they will more likely reduce inflammation due to the presence of the carotenoids, lutein and zeaxanthin that are highly available in eggs.

In this study, the investigators are evaluating three main things

* Atherogenic dyslipidemia by measuring plasma lipids and lipoprotein mean size and subfractions by nuclear magnetic resonance.
* Glucose metabolism by measuring plasma glucose, insulin, insulin resistance and glycosylated hemoglobin.
* Inflammation by measuring liver enzymes, C reactive protein, tumor necrosis factor-alpha, interleukin-6.

All these measurements were done 24 weeks after completion of the study All data will be presented 1 year after completion of the study

ELIGIBILITY:
Inclusion Criteria:

* diabetic subjects diagnosed by physician
* male and female
* 35-65 years
* Glycosylated hemoglobin < 9%

Exclusion Criteria:

* taking ezetimibe
* heart disease
* renal problems
* cancer
* thyroid problems

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
glycosylated hemoglobin | Assessed at base line and at the end of 5 weeks after the consumption of eggs and at the end of 5 weeks after the consumption of oatmeal
  Glycosylated hemoglobin had to be < 9% as one of the inclusion criteria. This parameter was assessed after 5 weeks that the subjects consumed the egg and after 5 weeks after the subjects were consuming the oatmeal.

SECONDARY OUTCOMES:
plasma LDL cholesterol | Measured at baseline and 5 weeks after the consuming the eggs and 5 weeks after consuming the oatmeal
  This parameter was assessed to ensure that no significant changes in LDL cholesterol occurred by egg intake or oatmeal intake. LDL cholesterol was assessed after 5 weeks of consuming the eggs and 5 weeks of consuming the oatmeal.

OTHER OUTCOMES:
tumor necrosis factor alpha | Assessed after 5 weeks of consuming the eggs and after 5 weeks of consuming the oatmeal
  This parameter was measured to determine whether egg intake favorably would affect inflammation in diabetic subjects. Tumor necrosis factor alpha was measured after 5 weeks of consuming the eggs and 5 weeks after consuming the oatmeal.

CONTACTS AND LOCATIONS:
Overall Officials: Maria-Luz Fernandez, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Centro de Investigacion y Desarrollo, Hermosillo, Sonora, Mexico